CLINICAL TRIAL: NCT03546881
Title: A Prospective Single Center Randomized Interventional Controlled Open Trial Comparing Patient and Staff Safety During Peripheral Endovascular Arterial Revascularisation Using Advanced Imaging Guidance Technology to Control Group Without Imaging Guidance.
Brief Title: Safety of Fusion Guidance During Peripheral Revascularisation
Acronym: SOFtPERIPHERAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination of the research following an internal reorganization of the team no longer allowing the necessary resources to continue the study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC17_0473
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Arteriopathy
Keywords: PAOD; endovascular; fusion; radiation; exposure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm with fusion imaging guidance technology (Experimental): arm with fusion imaging guidance technology to perform the endovascular surgery, in addition to the traditional 2D X-ray screen system.
  Interventions: Procedure: fusion imaging guidance technology; Procedure: 2D X-ray screen
- Arm without fusion imaging guidance technology (Active Comparator): arm without fusion imaging guidance technology, using the traditional 2D X-ray screen system, to perform the endovascular surgery.
  Interventions: Procedure: 2D X-ray screen

INTERVENTIONS:
Procedure: fusion imaging guidance technology — Imaging fusion guidance overlay used during PAOD endovascular revascularisation
  Arms: Arm with fusion imaging guidance technology
Procedure: 2D X-ray screen — 2D X-ray screen during PAOD endovascular revascularisation

SUMMARY:
Study the Patient and staff Safety regarding the radiation exposure during the procedure with and without the fusion imaging guidance technology in treatment of peripheral artery disease.

DETAILED DESCRIPTION:
The investigators are proposing a prospective, monocentric trial to assess the use of fusion imaging in peripheral endovascular revascularisation. The main aim of this research is to prove that using fusion imaging guidance during peripheral endovascular revascularisation improve the patient and staff safety in the theatre, through a reduction of radiation exposure.

Peripheral artery occlusive disease (PAOD) is a worldwide well known disease, with atherosclerosis as a leading cause. One third of patients with PAOD are symptomatic, typically presenting with claudication, and in a very much less proportion with critical limb ischemia. These last patients are high risk for major limb amputation without revascularisation. Once symptomatic PAOD diagnosed, a CT-scan is required to assess the anatomy and if indicated an endovascular revascularisation of the lower limbs arteries is performed. This minimally invasive procedure allows the improvement of the hemodynamic flow into the lower limb, by positioning one or several stents inside the diseased arteries through a femoral or an humeral access under live X-rays (fluoroscopy) guidance.

X-rays are good at showing bones and radio-opaque endovascular tools, but they do not show soft tissues like the arteries, and they produce flat (2D) images that superimpose all the 3D anatomical features. In order to see the arteries, physicians have to inject iodinated contrast during high quality imaging recording, which can be toxic for the kidneys, and increases the amount of radiation used. Consequently, the drawbacks of this mini-invasive procedure are the X-rays radiation exposure for both patients and medical staff, and the need of iodinated contrast injection that can lead to lifelong kidney problems. Reducing both in order to decrease their respective toxicities must be a priority for the endovascular therapist. Several studies including guidelines recall basic safety standards for protection against X-rays and iodinated contrast exposure.

One way to reduce both radiation and contrast use is to improve clinicians' perception of intraoperative 3D vascular anatomy. Advanced imaging techniques allow overlay of a 3D version of the aorta from a pre-operative CT scan (a 3D vascular mask) onto the live X-ray image creating a '3D roadmap' - a virtual reality that helps guide surgery. It has been proven that using fusion imaging guidance during aortic endovascular repair reduce both contrast and radiation dose, especially if the registration protocol is contrast and almost radiation free. The investigators have recently completed research showing that they are able to use an advanced imaging application to dramatically reduce our radiation dose for complex aneurysms.

Traditionally, this advanced imaging application is currently available only in modern expensive hybrid theatres, and not used in everyday practice during peripheral endovascular revascularisation procedures. However new technologies are about to supply similar imaging to any interventional equipment, which will change the way endovascular procedures are performed worldwide. That's why using fusion imaging guidance routinely as a standard of care may be part of good practice to improve patient and staff safety. However, to our knowledge, the impact of using fusion on radiation dose and contrast use has not been validated for peripheral endovascular procedures.

This trial will examine the clinical benefits of using fusion imaging guidance during peripheral endovascular revascularisation procedures based on the radiation exposure, as compared with procedures without imaging guidance. The design of the study is to compare a prospective single centre cohort of 88 consecutive patients scheduled for an endovascular peripheral procedure and randomised either as using the imaging guidance overlay, or to a control cohort of patients whose procedure will be performed without imaging guidance (standard of care).

This study is a Low risk and constraints study, because it's a standard care procedure with no additional risks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Male or Female
* Aged 18 or older
* Have been scheduled for peripheral endovascular revascularisation of an occlusive arterial disease excluding isolated infra popliteal revascularisation
* Who have had a pre-operative diagnostic CT scan
* Able (in the investigator's opinion) and willing to comply with the study requirements
* Covered by the French public health insurance system

Exclusion Criteria:

* Female under the age of 50 years old.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Any patient requiring an associated procedure: renal or mesenteric angioplasty.
* Adult under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
DAP (Dose Aera Product in Gy.cm²) by the end of the procedure, | day 0, per procedure
  The DAP is a surrogate measurement for the entire amount of energy delivered to the patient by the beam.

SECONDARY OUTCOMES:
AK (Air Kerma, in Gy) | day 0, per procedure
  an indirect measurement automatically reported by the fluoroscopy equipment thus highly reproducible and responsive to change in X-rays emission
Number of DSA (Digital Subtraction Angiography) runs | day 0, per procedure
  runs (Digital subtraction angiography) along the procedure. The DSA allows high quality loop acquisition with subtraction of non-vascular structures that requires substantial additional radiation exposure compared with standard fluoroscopy
FT (Fluoroscopy Time, min). | day 0, per procedure
  a counting of the time spent using fluoroscopy.
Radiation exposure to the operator (Sv). | day 0, per procedure
  The operator's exposure to radiation, recorded by a live dosimeter
Iodinated contrast volume (ml). | day 0, per procedure
  repeated injections of contrast media contribute to the development of lifelong nephropathy, predominantly in patients with diabetic nephropathy (19.7%) and pre-existing renal impairment (3%-33%)
Total operative time ( min) | day 0, per procedure
  time of the operation, between the first puncture and the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Maurel, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Vascular surgery, Institut du Thorax, Nantes, France